CLINICAL TRIAL: NCT00780416
Title: A Phase 3 Study of MP-424 in Combination With Peginterferon Alfa-2b and Ribavirin, in Treatment-Naïve Subjects With Genotype 1 Hepatitis C
Brief Title: Efficacy and Safety of MP-424/Peginterferon Alfa-2b/Ribavirin Combination in Treatment-Naïve Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G060-A6
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Results first posted 2012-08-20 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Hepatitis C
Keywords: Chronic Hepatitis C; Protease Inhibitor; Telaprevir; Peginterferon Alfa-2b; Ribavirin
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — telaprevir; Ribavirin; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TRV/PEG/RBV (Experimental)
  Interventions: Drug: MP-424; Drug: Ribavirin; Drug: Peginterferon Alfa-2b
- PEG/RBV (Active Comparator)
  Interventions: Drug: Ribavirin; Drug: Peginterferon Alfa-2b

INTERVENTIONS:
Drug: MP-424 — 750 mg every 8 hours for 12 weeks
  Other Names: Telaprevir
  Arms: TRV/PEG/RBV
Drug: Ribavirin — 600 - 1000 mg/day based on body weight for 24 weeks
Drug: Peginterferon Alfa-2b — 1.5 mcg/kg/week for 24 weeks
Drug: Ribavirin — 600 - 1000 mg/day based on body weight for 48 weeks
Drug: Peginterferon Alfa-2b — 1.5 mcg/kg/week for 48 weeks

SUMMARY:
This study will evaluate the efficacy and safety of MP-424 with Peginterferon Alfa-2b (PEG-IFN) and Ribavirin (RBV) in treatment-naïve patients with (Genotype 1) hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* Genotype 1, chronic hepatitis C
* Treatment-naïve (patient who has received no previous interferon based treatment for hepatitis C)
* Able and willing to follow contraception requirements

Exclusion Criteria:

* Cirrhosis of the liver or hepatic failure
* Hepatitis B surface antigen-positive or HIV antibodies-positive
* History of, or concurrent hepatocellular carcinoma
* History of, or concurrent depression, schizophrenia; or suicide attempt in the past
* Pregnant, lactating, or suspected pregnant patients, or male patients whose female partner is pregnant

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2008-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fumitaka Suzuki, MD, Principal Investigator — Department of Hepatology, Toranomon Hospital
Locations (1):
- Toranomon Hospital, Kawasaki, Takatsu-ku, Japan

REFERENCES:
- [Result] Kumada H, Toyota J, Okanoue T, Chayama K, Tsubouchi H, Hayashi N. Telaprevir with peginterferon and ribavirin for treatment-naive patients chronically infected with HCV of genotype 1 in Japan. J Hepatol. 2012 Jan;56(1):78-84. doi: 10.1016/j.jhep.2011.07.016. Epub 2011 Aug 7. PMID 21827730

RESULTS

PARTICIPANT FLOW:
Groups:
- TRV/PEG/RBV: Drug: MP-424 750 mg every 8 hours for 12 weeks Other Name: Telaprevir
  Drug: Ribavirin 600 - 1000 mg/day based on body weight for 24 weeks
  Drug: Peginterferon Alfa-2b 1.5 mcg/kg/week for 24 weeks
- PEG/RBV: Drug: Ribavirin 600 - 1000 mg/day based on body weight for 48 weeks
  Drug: Peginterferon Alfa-2b 1.5 mcg/kg/week for 48 weeks
Period: Overall Study
Arm/Group | TRV/PEG/RBV | PEG/RBV
Started | 126 | 63
Completed | 114 | 54
Not Completed | 12 | 9
Not completed — Physician Decision | 3 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TRV/PEG/RBV | PEG/RBV | Total
Number analyzed (Participants) | 126 | 63 | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (10.4) | 52.2 (9.7) | 51.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 30 | 90
  Male | 66 | 33 | 99

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Achieving Undetectable Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) at 24 Weeks After Completion of Drug Administration (SVR, Sustained Viral Response)
Time Frame: After 24 weeks of follow-up
Measure: Number (95% Confidence Interval); unit: percentage of subjects achieving SVR
Arm/Group | TRV/PEG/RBV | PEG/RBV
Number analyzed (Participants) | 126 | 63
percentage of subjects achieving SVR | 73.0 [64.4 to 80.5] | 49.2 [36.4 to 62.1]

ADVERSE EVENTS:
Arm/Group | TRV/PEG/RBV | PEG/RBV
Serious Adverse Events (participants affected / at risk) | 15/126 | 6/63
Other Adverse Events (participants affected / at risk) | 126/126 | 63/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TRV/PEG/RBV (N=126) | PEG/RBV (N=63)
Gastroenteritis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Mania (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Anisometropia (Eye disorders) | 0 | 1
Macular hole (Eye disorders) | 0 | 1
Retinoschisis (Eye disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Drug rash with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TRV/PEG/RBV (N=126) | PEG/RBV (N=63)
Nasopharyngitis (Infections and infestations) | 23 | 18
Anaemia (Blood and lymphatic system disorders) | 113 | 46
Decreased appetite (Metabolism and nutrition disorders) | 41 | 16
Hyperuricaemia (Metabolism and nutrition disorders) | 20 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 8 | 0
Insomnia (Psychiatric disorders) | 40 | 17
Headache (Nervous system disorders) | 48 | 32
Dysgeusia (Nervous system disorders) | 34 | 10
Dizziness (Nervous system disorders) | 12 | 7
Hypoaesthesia (Nervous system disorders) | 10 | 1
Retinopathy (Eye disorders) | 11 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 6
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Diarrhoea (Gastrointestinal disorders) | 34 | 19
Vomiting (Gastrointestinal disorders) | 37 | 9
Nausea (Gastrointestinal disorders) | 32 | 7
Abdominal discomfort (Gastrointestinal disorders) | 23 | 12
Stomatitis (Gastrointestinal disorders) | 24 | 12
Constipation (Gastrointestinal disorders) | 14 | 13
Abdominal pain upper (Gastrointestinal disorders) | 8 | 7
Haemorrhoids (Gastrointestinal disorders) | 7 | 2
Cheilitis (Gastrointestinal disorders) | 5 | 5
Rash (Skin and subcutaneous tissue disorders) | 48 | 18
Alopecia (Skin and subcutaneous tissue disorders) | 51 | 29
Drug eruption (Skin and subcutaneous tissue disorders) | 37 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 23 | 13
Pruritus generalised (Skin and subcutaneous tissue disorders) | 9 | 2
Erythema (Skin and subcutaneous tissue disorders) | 9 | 13
Eczema (Skin and subcutaneous tissue disorders) | 8 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 3
Pyrexia (General disorders) | 98 | 46
Malaise (General disorders) | 73 | 30
Injection site erythema (General disorders) | 33 | 21
Injection site reaction (General disorders) | 29 | 16
Influenza like illness (General disorders) | 22 | 16
Thirst (General disorders) | 7 | 1
White blood cell count decreased (Investigations) | 86 | 46
Platelet count decreased (Investigations) | 81 | 23
Blood uric acid increased (Investigations) | 65 | 5
Hyaluronic acid increased (Investigations) | 64 | 25
Blood creatinine increased (Investigations) | 32 | 0
Blood bilirubin increased (Investigations) | 22 | 13
Blood triglycerides increased (Investigations) | 36 | 11
Blood phosphorus decreased (Investigations) | 16 | 13
Neutrophil count decreased (Investigations) | 18 | 9
Blood potassium decreased (Investigations) | 12 | 2
Blood pressure increased (Investigations) | 10 | 2
High density lipoprotein decreased (Investigations) | 8 | 9
Protein total decreased (Investigations) | 7 | 3
Blood thyroid stimulating hormone decreased (Investigations) | 4 | 5
Contusion (Injury, poisoning and procedural complications) | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other